CLINICAL TRIAL: NCT00002097
Title: A Phase I/II Clinical Study of Nystatin I.V. (Intravenous) in Patients With HIV Infection.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Argus Pharmaceuticals (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 103B; AR-91-35,606-004
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1994-04

CONDITIONS: HIV Infections
Keywords: Nystatin; Acquired Immunodeficiency Syndrome; AIDS-Related Complex
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Nystatin

INTERVENTIONS:
Drug: Nystatin

SUMMARY:
To evaluate the clinical toxicity, safety, and maximum tolerated dose (MTD) of intravenous nystatin in patients with HIV infection. To evaluate the potential anti-HIV activity and clinical pharmacology of intravenous nystatin.

DETAILED DESCRIPTION:
Cohorts of three patients each are treated at escalating doses of intravenous nystatin, administered every other day, until the MTD is reached. Each cohort is observed for toxicity for at least 2 weeks before escalation in subsequent patient cohorts is initiated.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Required:

* Aerosolized pentamidine (300 mg once a month) for PCP prophylaxis in patients with CD4 count <= 200 cells/mm3. (Patients with CD4 count > 200 cells/mm3 who are already on aerosolized pentamidine may continue such therapy at the discretion of the investigator.)

Allowed:

* Prophylaxis against Mycobacterium avium Complex in patients with CD4 count <= 100 cells/mm3.

Concurrent Treatment:

Allowed:

* Local treatment for Kaposi's sarcoma lesions with less than 25 percent increase in measurable disease.

Patients must have:

* HIV antibody positivity.
* Absolute CD4 count < 500 cells/mm3 on two determinations within 15 days prior to study entry.
* At least 6 months of prior zidovudine (AZT) therapy.
* No active opportunistic infection requiring ongoing therapy.
* Normal neurologic status by standard assessment.
* Life expectancy of at least 6 months.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms and conditions are excluded:

* Neoplasm other than basal cell carcinoma of the skin or stable untreated HIV-related Kaposi's sarcoma (provided there is no progression in the Kaposi's sarcoma beyond 25 percent of measurable disease).
* Clinically significant cardiac disease.
* Known hypersensitivity to polyene antibiotics.

Patients with the following prior conditions are excluded:

* History of myocardial infarction or arrhythmias.

Prior Medication:

Excluded within 2 weeks prior to study entry:

* Antiretroviral agents or interferons.
* Biological response modifiers.
* Corticosteroids.
* Cytotoxic chemotherapeutic agents.
* Drugs that can cause neutropenia or significant nephrotoxicity.
* Rifampin or rifampin derivatives.
* Systemic anti-infectives.

Prior Treatment:

Excluded within 2 weeks prior to study entry:

* Radiation therapy. Active drug or alcohol abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Twelve Oaks Hosp, Houston, Texas, United States

REFERENCES:
- [Background] Rios A, Brewton G, Crofoot G, Quesada J, Lenk R, Lopez-Berenstein G. A phase I-II clinical study of Nystatin-LF IV in patients with HIV infections. Int Conf AIDS. 1993 Jun 6-11;9(1):483 (abstract no PO-B26-2089)